CLINICAL TRIAL: NCT06440629
Title: A Multi-center, Open, Randomized, 18-month, Parallel-group, Superiority Study to Compare the Effect of Proactive Therapeutic Drug Monitoring Versus Standard of Care With Regards to Maintenance of Sustained Disease Control Without Flare in Adults With Rheumatoid Arthritis Treated With a Subcutaneous Tumor Necrosis Factor Inhibitor
Brief Title: Effect of Proactive Therapeutic Drug Monitoring on Maintenance of Sustained Disease Control in Adults With Rheumatoid Arthritis on a Subcutaneous TNF Inhibitor: The Rheumatoid Arthritis Therapeutic DRUg Monitoring Trial (RA-DRUM)
Acronym: RA-DRUM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Oslo University Hospital (Other); Karolinska University Hospital (Other); Queen Mary University of London (Other); Medical University of Vienna (Other); Alesund Hospital (Other); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); Drammen sykehus (Other); University Hospital of North Norway (Other); Førde Hospital Trust (Other); Hospital of Southern Norway Trust (Other); Haukeland University Hospital (Other); Ostfold Hospital Trust (Other); Lillehammer Hospital for Rheumatic Diseases (Other); Vestre Viken Hospital Trust (Other); Haugesund Rheumatism Hospital (Other); Betanien Hospital (Other); Helgeland Hospital Trust (Other); Nordlandssykehuset HF (Other); Carol Davila University of Medicine and Pharmacy (Other); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU CT No 2023-510184-35-00
Record Dates: First submitted 2024-05-23; First posted 2024-06-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Therapeutic drug monitoring; Tumor necrosis factor inhibitor
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Masking Description: The joint assessor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TDM-group (Experimental): In the TDM-group, the TNFi dose will be adjusted in order to keep the drug level within the therapeutic range
  Interventions: Drug: Therapeutic drug monitoring (TDM) of adalimumab
- Standard of Care group (No Intervention): In the Standard of Care group, TNFi will be administered according to standard of care without knowledge of serum drug levels or ADAb

INTERVENTIONS:
Drug: Therapeutic drug monitoring (TDM) of adalimumab — In the TDM-group, the adalimumab dose will be adjusted according to the following algorithms in order to keep the drug level within the therapeutic range:
  * Serum drug level within therapeutic range : keep dose
  * Low drug levels, ADAb undetectable or low levels : Decrease dosing interval by one week to a maximum of 40 mg/week
  * Low drug levels, ADAb high levels : Switch to another therapy
  * High drug levels : Increase dosing interval by one week up to a maximum of 6 weeks
  Arms: TDM-group

SUMMARY:
The goal of this clinical trial is to compare therapeutic drug monitoring (TDM) versus Standard of care in patients with rheumatoid arthritis treated with a subcutaneous tumor necrosis factor inhibitor (adalimumab).

The main question it aims to answer is:

Is TDM superior to standard of care in order to maintain sustained disease control without flares?

Participants will be followed with blood sampling every second month, measuring serum drug levels and anti-drug antibodies of the TNFi. In the TDM-group, the researchers will adjust the dosage of the TNFi based on knowledge on optimal therapeutic ranges. In the Standard of care group, the TNFi will be administered according to standard of care without knowledge of serum drug levels or anti-drug antibodies.

DETAILED DESCRIPTION:
There is a considerable variation in serum drug levels among rheumatoid arthritis (RA) patients on tumor necrosis factor inhibitors (TNFi), and a high number develop neutralizing anti-drug antibodies (ADAb). Sub-therapeutic drug levels and ADAb formation are major contributors to TNFi treatment failure and disease flare. Proactive therapeutic drug monitoring (TDM), i.e., individualized drug dosing based on regular assessments of serum drug levels and ADAb, has the potential to optimize the efficacy and safety of TNFi treatment.

The aim of the RA-DRUM trial is to assess whether TDM is superior to standard of care in order to maintain sustained disease control without flares in patients with RA treated with the SC TNFi adalimumab.

Participants will be randomized to:

* Administration of TNFi based on proactive TDM (TDM group)
* Administration of TNFi based on standard of care without knowledge of serum drug levels or ADAb status (Standard of care group)

Participants will be followed for 18 months with on-site visits at baseline, 4, 8, 12 and 18 months and digital visits at 2, 6, 10, 14, and 16 months. Blood sampling for serum drug levels and anti-drug antibodies will be done at all visits.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of RA
2. ≥ 18 and under 75 years of age at screening
3. On stable therapy with standard dose of a SC TNFi (adalimumab) for a minimum of 3 months and a maximum of 24 months
4. In low disease activity or remission (DAS28-CRP under 3.2) and indication for continuation of treatment according to the treating physician
5. Subject capable of understanding and signing an informed consent form

Exclusion Criteria:

1. Major comorbidities, such as previous malignancies within the last 5 years, uncontrolled diabetes mellitus, severe infections (including HIV), uncontrollable hypertension, severe cardiovascular disease (NYHA class 3 or 4), severe respiratory diseases, demyelinating disease, significant chronic widespread pain syndrome, significant renal or hepatic disease, and/or other diseases or conditions which either contraindicate treatment with SC TNFi or make adherence to the protocol difficult
2. Hypersensitivity to sc TNFi (adalimumab).
3. Pregnancy, or subject considering becoming pregnant during the study period
4. Psychiatric or mental disorders, alcohol abuse or other substance abuse, language barriers, or other factors that makes adherence to the study protocol difficult
5. Changes in csDMARD co-medication, including dose changes of csDMARD or changes in the dose of corticosteroids within the last 2 months
6. Co-medication with bDMARD, tsDMARD, or other immunosuppressive drugs (excluding csDMARD and corticosteroids ≤ 7.5 mg prednisolone (or equivalent) once daily).
7. Active participation in any other interventional study.
8. In need of live vaccines during the study period.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained disease control over the follow-up period of 18 months without flare | 4, 8, 12, 18 months
  A flare defined as either of the following:
  A combination of an increase in Disease Activity Score using 28 joints C-reactive protein (DAS28-CRP) ≥ 1.2, or ≥ 0.6 if DAS28-CRP ≥ 3.2, AND ≥ 2 swollen joints on examination of 44 joints
  OR
  Consensus between patient and physician that a disease flare has occurred, leading to a major change* in treatment
  *Please see protocol for the definition of a major change in treatment (due to word restrictions)

SECONDARY OUTCOMES:
Disease activity assessed by Disease Activity Score using 28 joints C-reactive protein (DAS28-CRP) | 4, 8, 12, and 18 months
  The DAS28-CRP composite score includes the 28 tender and swollen joint counts, CRP and a Patient Global Assessment of Disease activity (PGA).
  The DAS28-CRP is calculated as follows:
  DAS28-CRP = 0.56*√ (tender joints 28) + 0.28*√ (swollen joints 28) + 0.36*ln(CRP (mg/L)+1) + 0.014*PGA + 0.96 High disease activity is defined as a DAS28-CRP value > 5.1, moderate disease activity as DAS28-CRP > 3.2 - 5.1, low disease activity as a DAS28-CRP-value of 2.6 - 3.2, and remission as DAS28-CRP < 2.6
  PGA is measured on a 100 mm VAS according to the question: "Considering all the ways your arthritis has affected you, how did you feel your arthritis was over the last week?" (on a 0-100mm Visual Analogue Scale (VAS) with with 0 = excellent and 100 = very poor).
Disease activity measured by 44 joint count | 4, 8, 12, and 18 months
  44 joint count are included in the original Disease Activity Score (DAS) and in addition to the joints included in DAS28 it includes the MTP joints and the sternoclavicular joints for a more comprehensive valuation of the participants' joints.
Patient Global assessment of disease activity (PGA) | 4, 8, 12, and 18 months
  PGA is measured on a 100 mm VAS according to the question: "Considering all the ways your arthritis has affected you, how did you feel your arthritis was over the last week?" (on a 0-100mm Visual Analogue Scale (VAS) with with 0 = excellent and 100 = very poor).
Evaluators Global Assessment of Disease Activity (EGA) | 4, 8, 12, and 18 months
  EGA is measured on a NRS according to the question "Please rate the patient's overall (global) disease activity", with 0 = best and 10 = worst.
Disease activity assessed by Clinical Disease Activity Index (CDAI) | 4, 8, 12, and 18 months
  CDAI includes the 28 tender and swollen joint counts, Patient Global Assessment of Disease activity (PGA) and Evaluators Global Assessment of Disease Activity (EGA)
  The formula for CDAI is: swollen joints 28 + tender joints 28 + (PGA (VAS 0-100)/10) + EGA (NRS 0-10).
  PGA is measured on a 100 mm VAS according to the question: "Considering all the ways your arthritis has affected you, how did you feel your arthritis was over the last week?" (on a 0-100mm Visual Analogue Scale (VAS) with with 0 = excellent and 100 = very poor).
  EGA is measured on a NRS according to the question "Please rate the patient's overall (global) disease activity", with 0 = best and 10 = worst.
Disease activity assessed by Simple Disease Activity Index (SDAI) | 4, 8, 12, and 18 months
  SDAI includes the 28 tender and swollen joint counts, Patient Global Assessment of Disease activity (PGA) and Evaluators Global Assessment of Disease Activity (EGA) and C-reactive protein (CRP).
  The formula for SDAI is: swollen joints 28 + tender joints 28 + (PGA(VAS 0-100)/10) + EGA(NRS 0-10) + (CRP (mg/dL)/10).
  PGA is measured on a 100 mm VAS according to the question: "Considering all the ways your arthritis has affected you, how did you feel your arthritis was over the last week?" (on a 0-100mm Visual Analogue Scale (VAS) with with 0 = excellent and 100 = very poor).
  EGA is measured on a NRS according to the question "Please rate the patient's overall (global) disease activity", with 0 = best and 10 = worst.
Remission assessed by American College of Rheumatology (ACR)/European Alliance of Associations for Rheumatology (EULAR) remission criteria | 4, 8, 12, and 18 months
  The ACR/EULAR remission criteria defines a patient in remission when either
  1. the patient is in Boolean 2.0 remission with each of the variables tender joint count, swollen joint count and CRP having a value of ≤1 and Patient Global Assessment of Disease activity (PGA) having a value ≤ 2 (PGA on a Visual Analogue Scale (VAS)100mm/10 with 0=best and 100= worst, CRP in mg/dl) OR
  2. the SDAI score is ≤ 3.3
Rheumatoid Arthritis Impact of Disease (RAID) | 4, 8, 12, and 18 months
  The RAID questionnaire includes seven domains with the following relative weights: pain (0.21), functional disability (0.16), fatigue (0.15), emotional well-being (0.12), sleep (0.12), coping (0.12) and physical well-being (0.12) each rated on an Numeric Rating Scale (NRS) (0-10 with 0=best and 10=worst). The rates of each domain are weighted and summed to form a score in the range of 0-10
Evaluation of physical function measured by Modified Health Assessment Questionnaire (MHAQ) | 4, 8, 12, and 18 months
  The MHAQ includes eight items covering the physical function of patients with inflammatory joint diseases.
  Each item is scored on a categorical 0-3 scale (0=best and 3= worst) and the sum score is divided by 8 to form the MHAQ score 0.0 to 3.0
Number and type of adverse events (AE) | 4, 8, 12, and 18 months
  Assessments of AE
Drug survival | 4, 8, 12, and 18 months
  Drug survival assessed by survival analyses
Drug consumption | 18 months
  Assessments of drug consumption
Occurrence of anti-drug antibodies (ADAb) | 2, 4, 6, 8, 10, 12, 14, 16, 18 months
  ADAb will be assessed in all serum samples with adalimumab levels <3mg/L.
Serum drug levels | 2, 4, 6, 8, 10, 12, 14, 16, 18 months
  Serum drug levels will be assessed at all visits, both clinical and digital.

OTHER OUTCOMES:
European Quality of Life 5 Dimensions (EQ-5D) | 2, 4, 6, 8, 10, 12, 14, 16, 18 months
  The EQ-5D is a utility instrument for measurement of health-related quality of life.
  It consists of 5 dimensions. Each dimension is scored on a level from 1 to 5:
  LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme
  The health state is referred to by a 5-digit code, e.g. state 11111 indicates no problems on any of the five dimensions, while state 55555 indicate extreme problems on all of the five dimensions.
36-Item Short-form health survey (SF-36) | 2, 4, 6, 8, 10, 12, 14, 16, 18 months
  The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8- scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index (SF-6D). It is a generic measure, as opposed to one that targets a specific age, disease, or treatment group. Accordingly, the SF-36 has proven useful in surveys of general and specific populations, comparing the relative burden of diseases, and in differentiating the health benefits produced by a wide range of different treatments.
Work Productivity and Activity Impairment Questionnaire: Rheumatoid Arthritis (WPAI:RA) | 2, 4, 6, 8, 10, 12, 14, 16, 18 months
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a tool that assesses impairments in both work and daily activities. It consists of six items that determine employment status and measure absenteeism caused by health issues, presenteeism, and overall health-related impairment in both paid work and regular activities over the preceding 7 days. The questionnaire yields four outcomes: i) the percentage of work time missed due to health; ii) the percentage of impairment experienced while working due to health in the past 7 days; iii) the percentage of overall work impairment; iv) activity impairment resulting from health issues. Participants will be asked to answer the Work Productivity and Activity Impairment Questionnaire: Rheumatoid Arthritis V2.0.
Rheumatoid arthritis flare questionnaire (RA-FQ) | 2, 4, 6, 8, 10, 12, 14, 16, 18 months
  The RA-FQ was developed by the Omeract group to identify and measure flares in patients with RA. It encompasses pain, physical impairment, fatigue, stiffness, and participation, and the score is calculated as the sum of responses for the 5 items (maximum 50).
Adherence | 2, 4, 6, 8, 10, 12, 14, 16, 18 months
  At each visit (every two months), the participant will fill out a questionnaire assessing compliance in into the eCRF.
Co-medication | 4, 8, 12, and 18 months
  Registration of co-medication will be made at each clinical visit.
Consentration of C-reactive protein (CRP) | 4, 8, 12, and 18 months
  C-reactive protein (CRP) will be measured at all clinical visits.
Erythrocyte sedimentation rate (ESR) | 4, 8, 12, and 18 months
  Erythrocyte sedimentation rate (ESR) will be measured at all clinical visits.

CONTACTS AND LOCATIONS:
Overall Officials: Espen A Haavardsholm, Phd, MD, Study Director — Diakonhjemmet Hospital
Locations (22):
- Medical University Vienna, Vienna, Austria
- Humanitas Research Hospital, Milan, Italy
- Norway (16):
  - Diakonhjemmet sykehus, Oslo, N-0319
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Nordland Hospital Trust, Bodø
  - Drammen Hospital, Drammen
  - Førde Hospital Trust, Førde
  - Haugesund Rheumatism Hospital, Haugesund
  - Hospital of Southern Norway Trust, Kristiansand
  - Lillehammer Hospital for Rheumatic Diseases, Lillehammer
  - Helgeland Hospital Trust, Mo i Rana
  - Østfold Hospital Trust, Moss
  - Martina Hansen's Hospital, Sandvika
  - Betanien Hospital, Skien
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St.Olavs Hospital, Trondheim
- Carol Davila University of Medicine and Pharmacy Bucharest, Bucharest, Romania
- Sweden (2):
  - Sahlgrenska Universitetssjukehuset, Gothenburg
  - Karolinska University Hospital, Stockholm
- Queen Mary, London, SW15 5PN, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
A de-identified patient data set can be made available to researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 10 years after publishing
Access Criteria: The data will only be made available after submission of a project plan outlining the reason for the request and any proposed analyses, and will have to be approved by the RA-DRUM steering group. Project proposals can be submitted to the corresponding author. Data sharing will have to follow appropriate regulations.

DOCUMENTS (1):
  • Study Protocol (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT06440629/Prot_000.pdf